CLINICAL TRIAL: NCT05119907
Title: A Phase II Open Label Study of Sacituzumab Govitecan in Patients With Solid Tumor
Brief Title: Study of Sacituzumab Govitecan in Patients With Solid Tumor
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EVER-132-003; CTR20210912 (Registry Identifier: China: Drug Clinical Trial Registration and Information Disclosure Platform)
Record Dates: First submitted 2021-11-03; First posted 2021-11-15 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Solid Tumor
MeSH Terms: interventions — sacituzumab govitecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Cohort A: Esophageal Squamous Cell Carcinoma (ESCC) (Experimental): Participants will receive Sacituzumab Govitecan-hziy (SG) 8 or 10 mg/kg on Days 1 and 8 of a 21-day cycle. Participants will continue treatment until disease progression or intolerable toxicity or consent withdrawal for any reason.
  Interventions: Drug: Sacituzumab Govitecan-hziy
- Cohort B: Gastric or Gastroesophageal Junction Adenocarcinoma (G/GEJC) (Experimental): Participants will receive SG 8 or 10 mg/kg on Days 1 and 8 of a 21-day cycle. Participants will continue treatment until disease progression or intolerable toxicity or consent withdrawal for any reason.
  Interventions: Drug: Sacituzumab Govitecan-hziy
- Cohort C: Cervical Cancer (CC) (Experimental): Participants will receive SG 10 mg/kg on Days 1 and 8 of a 21-day cycle. Participants will continue treatment until disease progression or intolerable toxicity or consent withdrawal for any reason.
  Interventions: Drug: Sacituzumab Govitecan-hziy
- Cohort D: Biliary Tract Cancer (BTC) (Experimental): Participants will receive SG 8 or 10 mg/kg on Days 1 and 8 of a 21-day cycle. Participants will continue treatment until disease progression or intolerable toxicity or consent withdrawal for any reason.
  Interventions: Drug: Sacituzumab Govitecan-hziy
- Cohort E: Lung Adenocarcinoma (LAC) (Experimental): Participants will receive SG 10 mg/kg on Days 1 and 8 of a 21-day cycle. Participants will continue treatment until disease progression or intolerable toxicity or consent withdrawal for any reason.
  Interventions: Drug: Sacituzumab Govitecan-hziy

INTERVENTIONS:
Drug: Sacituzumab Govitecan-hziy — Administered intravenously
  Other Names: IMMU-132; Trodelvy™; GS-0132

SUMMARY:
The goal of this study is to see how effective the study drug, sacituzumab govitecan-hziy, is in participants with solid tumor.

ELIGIBILITY:
Key Inclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0 or 1.
* Histologically or cytologically-documented, incurable locally advanced or metastatic solid tumor of one of the following types:

  * Cohort A: oesophageal squamous-cell carcinoma that was refractory or intolerant to fluoropyrimidine-based, platinum-based, and taxane-based chemotherapy.
  * Cohort B: gastric adenocarcinoma that was refractory or intolerant to fluoropyrimidine-based, platinum-based, and taxane-based chemotherapy.
  * Cohort C: cervical cancer that was refractory or intolerant to platinum-based and taxane-based chemotherapy.
  * Cohort D: biliary tract cancer, including intrahepatic cholangiocarcinoma (IHCC), extrahepatic cholangiocarcinoma (EHCC), and gallbladder cancer (GBC), with exception of ampullary carcinoma, progressed during or after first line platinum-based or fluoropyrimidine-based chemotherapy.
  * Cohort E: lung adenocarcinoma with activating genomic alterations (EGFR/ ALK/ ROS1/ BRAF/ MET/ RET) that was refractory or intolerant to targeted tyrosine kinase inhibitors (TKIs) and had not received platinum-based chemotherapy for unresectable local advanced or metastatic disease, and no suitable or willing to receive platinum-based chemotherapy.
* Measurable disease by computed tomography (CT) or magnetic resonance imaging (MRI) in accordance with RECIST v 1.1, bone-only disease is not measurable and is not permitted.
* Availability of archival tumor tissue or newly acquired biopsy (unstaining tumor slides, recommended from metastasis sites).
* Adequate bone marrow, hepatic and renal function.
* Recovered from all prior treatment-related toxicities to Grade 1 or less by NCI-CTCAE v 5.0 (except alopecia or peripheral neuropathy that may be Grade 2 or less).
* Individuals must have completed all prior cancer treatments at least 2 weeks prior to the first dose including chemotherapy , radiotherapy and major surgery. Prior antibody treatment for cancer must have been completed at least 3 weeks prior to the first dose.
* Individuals must have at least a 3-month life expectancy.

Key Exclusion Criteria:

* Previous treatment with topoisomerase I inhibitors as a free form or as other formulations.
* Previous treatment with Trop-2 targeted therapy.
* Individuals with a history of or current central nervous system (CNS) metastases.
* Known additional malignancy within 3 years prior to enrollment with the exception of curatively treated basal cell carcinoma of the skin, squamous cell carcinoma of the skin and/or curatively resected in situ cancers.
* Individuals known to be human immunodeficiency virus positive.
* Individuals with active hepatitis B virus (HBV), or hepatitis C virus (HCV) infection. Hepatitis B core antibody (HBcAb) testing is required and if positive, then HBV DNA testing will be performed and if positive the individual will be excluded.
* Known history of unstable angina, myocardial infarction (MI), or chronic heart failure present within 6 months of first dose or clinically significant cardiac arrhythmia (other than stable atrial fibrillation) requiring anti-arrhythmia therapy or left ventricular ejection fraction < 50%.
* Known history of clinically significant active chronic obstructive pulmonary disease, or other moderate-to-severe chronic respiratory illness present within 6 months of the first dose.
* Infection requiring systematic antibiotic use within 1 week of the first dose.
* Individuals with active chronic inflammatory bowel disease (ulcerative colitis, Crohn disease) and individuals with a history of bowel obstruction or gastrointestinal (GI) perforation.
* High dose systemic corticosteroids within 2 weeks prior to the first dose (however, low dose corticosteroids ≤ 10 mg prednisone or equivalent daily are permitted provided the dose is stable for 4 weeks).
* Individuals who have received a live vaccine within 30 days of first dose.

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2021-10-12 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) According to Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v 1.1) By Investigator Assessment | Up to 4 years
  ORR is defined as the proportion of participants who achieve a complete response (CR) or partial response (PR).

SECONDARY OUTCOMES:
Duration of Response (DOR) | Up to 4 years
  DOR is defined as the time from the first documentation of CR or PR to the earlier of the first documentation of definitive progressive disease (PD) or death from any cause (whichever comes first).
Disease Control Rate (DCR) | Up to 4 years
  DCR is defined as the proportion of participants who achieve CR, PR, or stable disease (SD).
Progression-free Survival (PFS) | Up to 4 years
  PFS is defined as the time from the first dose of sacituzumab govitecan-hziy (SG) until the date of objective PD, or death (whichever comes first).
Overall Survival (OS) | Up to 4 years
  OS is defined as the time from the first dose of SG until death due to any cause.
Percentage of Participants Experiencing Adverse Events (AEs) According to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0 | First dose date up to 4 years plus 30 days
Percentage of Participants Experiencing Serious Adverse Events (SAEs) According to NCI CTCAE Version 5.0 | First dose date up to 4 years plus 30 days
Pharmacokinetic (PK) Parameter: Cmax of Sacituzumab Govitecan-hziy and Free SN-38 | Up to 4 years
  Cmax is defined as the maximum observed concentration of drug.
PK Parameter: Tmax of Sacituzumab Govitecan-hziy and Free SN-38 | Up to 4 years
  Tmax is defined as the time (observed time point) of Cmax.
PK Parameter: Ctrough of Sacituzumab Govitecan-hziy and Free SN-38 | Up to 4 years
  Ctrough is defined as the concentration of drug at the end of the dosing interval.
Percentage of Participants Who Developed Anti-Drug Antibodies (ADAs) Against SG | Up to 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (13):
- China (13):
  - Beijing Obstetrics and Gynecology Hospital, Capital Medical University, Beijing
  - Chinese Academy of Medical Sciences Cancer Hospital, Beijing
  - Beijing Cancer Hospital, Beijing
  - The First Hospital of Jilin University, Changchun
  - Fujian Cancer Hospital, Fuzhou
  - The Sixth Affiliated Hospital, Sun Yat-Sen University, Guangzhou
  - The First Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou
  - Zhejiang Cancer Hospital, Hangzhou
  - Harbin Medical University Cancer Hospital, Harbin
  - Anhui Provincial Hospital, Hefei
  - Jiangsu Province Hospital, Nanjing
  - Union Hospital Tongji Medical College Huazhong University of Science and Technology, Wuhan
  - Henan Cancer Hospital, Zhengzhou

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Gilead Clinical Trials Website — https://www.gileadclinicaltrials.com/study/?id=EVER-132-003